CLINICAL TRIAL: NCT03111927
Title: The Effect of Myelin-Relevant Nutrients in Infant Formula on Brain Myelination and Cognitive Development
Brief Title: Infant Nutrition and Brain Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16.14.NRC
Record Dates: First submitted 2017-02-28; First posted 2017-04-13 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Healthy; Infant Development
Keywords: Nutrition, Brain Development, Cognition, Heathy Infants
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: Multicenter, double blind, randomized, controlled, parallel group clinical trial, consisting of 2 arms randomized to receive either the investigational or the control product, and a nonrandomized, nonblinded arm of fully breastfed infants.
  3 groups: enriched level of myelin-relevant nutrients in an Infant Formula, standard level of myelin-relevant nutrients in an Infant Formula, breastfed infants
Who Masked: Participant, Investigator
Masking Description: Double blind - Infant Formula arms are blinded;
  * Reference Arm - unblinded epidemiological reference arm
  * Allocation: Randomized for formula arms, efficacy study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reference Arm: Breastfed (No Intervention): Epidemiological reference group of breastfed infants.
- Investigational (Experimental): Infant Formula: enriched level of myelin-relevant nutrients
  Interventions: Other: Infant Formula: enriched level of myelin-relevant nutrients
- Control (Active Comparator): Infant formula: standard level of myelin-relevant nutrients
  Interventions: Other: Infant formula: standard level of myelin-relevant nutrients

INTERVENTIONS:
Other: Infant Formula: enriched level of myelin-relevant nutrients — Feeding with the assigned infant formula begun as soon as the child was enrolled in the study (from 2 weeks up to 5 weeks of life) and lasted up to 12 months of age (+/- 2 weeks).
  The volume of feed required by the child per day depended upon age, weight, and appetite. The product was given daily ad libitum to the child from enrollment up to 12 months.
  Other Names: Infant Formula
  Arms: Investigational
Other: Infant formula: standard level of myelin-relevant nutrients — Feeding with the assigned infant formula begun as soon as the child was enrolled in the study (from 2 weeks up to 5 weeks of life) and lasted up to 12 months of age (+/- 2 weeks).
  The volume of feed required by the child per day depended upon age, weight, and appetite. The product was given daily ad libitum to the child from enrollment up to 12 months.
  Other Names: Infant Formula
  Arms: Control

SUMMARY:
Research study on the role of early life nutrition on brain and cognitive development during infancy and early childhood. Two blends of myelin-relevant nutrients at different levels were compared and a breastfed group was considered as epidemiological reference.

DETAILED DESCRIPTION:
This nutritional intervention study involved assessments in both the mother and her infant. The mother was asked to complete self-report questionnaires and to undergo a brief cognitive assessment. If the mother was not breastfeeding, a study product was provided and was consumed by the infant daily up to 12 months of life. The study also involved magnetic resonance imaging (MRI) brain scans of the infant's brain while asleep as well as evaluation of cognitive outcomes, including general cognitive development, and social-emotional development.

Once all trial subjects completed the 6-month timepoint (intervention part), an inferential statistical analysis of all data up to 6 months was performed.

Product codes (blinding) were broken to compare groups and an appropriate operational framework was put in place to maintain the individual assignment unknown to the Sponsor and Sites until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Term infants (≥ 37 weeks)
* Neuro typical development
* No major risk factors for learning, neurologic, or psychiatric disorder
* Between 2 weeks and maximum 5 weeks of age. If mother is breastfeeding she can choose the infant begin the trial prior 2 weeks.
* Parents/legal guardians willing and able to complete the informed consent process

Exclusion Criteria:

* Delayed birth (> 41 weeks gestation)
* Birth Weight < 2000 g or small for gestation age or large for gestational age
* Psychopharmacological treatment of mother using prohibited medications during pregnancy
* In utero exposure to alcohol abuse or illicit substances as per the American College of Obstetricians and Gynecologists
* Abnormalities on fetal ultrasound
* Complicated pregnancy
* Neonatal intensive care unit admission and/or emergency surgical delivery

Ages: 2 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Brain structural connectivity | 3, 6, 12, 18, and 24 months of life
  Longitudinal analysis de novo myelination and comparison between the 3 study arms De novo myelination being assessed by brain magnetic resonance imaging (MRI; multicomponent relaxometry). [Physiological marker, MRI].
Brain functional connectivity | 3, 6, 12, 18, and 24 months of life
  Cross-sectional analysis de novo myelination and comparison between the 3 study arms De novo myelination being assessed by brain magnetic resonance imaging (MRI; multicomponent relaxometry). [Physiological marker, MRI].
Brain De novo myelination | 3, 6, 12, 18, and 24 months of life
  Brain magnetic resonance imaging (MRI) derived measures (volumetric anatomical imaging) [Physiological marker, MRI].
Infant Cognitive Development | 6, 12, and 24 months of life
  Standardized neurodevelopment test.
Infant Early Learning Assessment | 18 and 24 months of life
  Computer-based cognitive tasks.
Infant Social Emotional Development | 3, 6, 12, 18, and 24 months of life
  Parent report questionnaire.

SECONDARY OUTCOMES:
Infant dietary assessment | 6, 9, 12, 18, and 24 months of life
  Three days food records are planned at the specified time-frames.
Breast milk nutrients profile | week 3, week 6, and 3 months of life
  Nutrients (vitamins, minerals, and other nutrients) levels analyses in breast milk nutrients (subsample) [Physiological parameter].
Brain structure | 3, 6, 12, 18, and 24 months of life
  MRI
Blood nutrients profile (optional) | 6, 12, and 24 months of life
  Nutrients (vitamins, minerals, and other nutrients) levels
Sleep | 3, 6, 12, 18, and 24 months of life
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sean Deoni, PhD, Principal Investigator — Rhode Island Hospital; Viren D'Sa, MD, Study Director — Rhode Island Hospital
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
MRI scans will be shared between sites. No Personal Identifiable Information will be shared.

REFERENCES:
- [Derived] Schneider N, Bruchhage MMK, O'Neill BV, Hartweg M, Tanguy J, Steiner P, Mutungi G, O'Regan J, Mcsweeney S, D'Sa V, Deoni SCL. A Nutrient Formulation Affects Developmental Myelination in Term Infants: A Randomized Clinical Trial. Front Nutr. 2022 Feb 10;9:823893. doi: 10.3389/fnut.2022.823893. eCollection 2022. PMID 35242798